CLINICAL TRIAL: NCT07186907
Title: Hydrocolloid Dressing for Diaper Dermatitis in NICU Hospitalized Neonates and Young Infants: A Quasi-Experimental Study
Brief Title: Hydrocolloid Dressings in Diaper Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gozde AKSUCU (Other)
Responsible Party: Sponsor-Investigator, Gozde AKSUCU, Assistant Professor (PhD), University of Beykent
Organization: University of Beykent (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-15-12
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diaper Dermatitis; Diaper Dermatitis Healing; Diaper Rash
Keywords: diaper dermatitis; hydrocolloid dressing; zinc oxide; NICU; quasi-experimental
MeSH Terms: conditions — Diaper Rash | interventions — Bandages, Hydrocolloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrocolloid dressing (Experimental)
  Interventions: Device: Hydrocolloid dressing
- Zinc oxide cream (Control group) (Active Comparator)
  Interventions: Drug: Zinc oxide cream %40

INTERVENTIONS:
Device: Hydrocolloid dressing — Hydrocolloid dressing was used for diaper dermatitis
  Arms: Hydrocolloid dressing
Drug: Zinc oxide cream %40 — Zinc oxide cream was used in diaper dermatitis.
  Arms: Zinc oxide cream (Control group)

SUMMARY:
Diaper dermatitis (commonly known as diaper rash) is one of the most frequent skin problems in newborns and infants, especially in neonatal intensive care units (NICUs). This study was designed to compare two treatment approaches for diaper dermatitis: hydrocolloid dressings and a cream containing 40% zinc oxide. The severity of diaper rash was evaluated at the beginning of treatment and at 24, 48, and 72 hours of follow-up.

DETAILED DESCRIPTION:
Diaper dermatitis (diaper rash) is a common skin problem in neonates and infants, often associated with prolonged exposure of the skin to moisture, urine, and stool. Infants hospitalized in neonatal intensive care units (NICUs) are particularly vulnerable due to frequent stools, immature skin, and exposure to irritants. This study was conducted to evaluate the effectiveness of hydrocolloid dressings compared with standard barrier cream containing 40% zinc oxide in the management of diaper dermatitis. A total of 44 infants hospitalized in a NICU and clinically diagnosed with diaper dermatitis were included. Infants were allocated into two groups: the intervention group received hydrocolloid dressings applied to the affected area, while the control group received zinc oxide cream. The severity of diaper dermatitis was assessed using a standardized clinical evaluation scale at baseline and at 24, 48, and 72 hours after initiation of the intervention. The primary aim was to compare changes in severity scores and healing time between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the NICU
* Body weight greater than 1000 g at the start of the intervention
* Gestational age above 26 weeks
* Diaper dermatitis diagnosis confirmed by a clinician
* Clinically stable condition at enrollment
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Congenital skin anomalies
* Dermatitis due to other dermatological conditions
* Systemic bacterial or fungal infections
* Receiving immunosuppressive treatment

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-17 (Actual)

PRIMARY OUTCOMES:
Change in diaper dermatitis severity score | Baseline, 24 hours, 48 hours, and 72 hours after initiation of intervention.
  The severity of diaper dermatitis will be assessed using the Clinical Evaluation Scale for Characterization of the Severity of Diaper Dermatitis (Stamatas & Tierney, 2014). Scores range from 0 (no dermatitis) to 3.0 (severe dermatitis), with 0.5-point increments. Higher scores indicate greater severity.
Time to complete healing of diaper dermatitis | Within 72 hours after initiation of intervention.
  Complete healing is defined as a diaper dermatitis score of "0" on the Clinical Evaluation Scale. The proportion of infants achieving complete healing within 72 hours will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol